CLINICAL TRIAL: NCT06918535
Title: Progressive Muscle Relaxation Vs Muscle Energy Technique on Nonspecific Neck Pain in Prolonged Computer Users. A Randomized Controlled Trial
Brief Title: Progressive Muscle Relaxation Vs Muscle Energy Technique on Nonspecific Neck Pain in Prolonged Computer Users.
Acronym: RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IQRA University (Other)
Collaborators: Dow University of Health Sciences (Other); Sindh Institute of Physical Medicine and Rehabilitation (Other)
Responsible Party: Principal Investigator, Syeda Waniya Riaz, Principal Investigator, IQRA University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IQRAU
Record Dates: First submitted 2025-03-18; First posted 2025-04-09 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Neck Pain; Chronic Neck Pain
Keywords: chronic pain; Computer user; Muscle relaxation; Progressive muscle relaxation,; neck pain; chronic neck pain; Sternocleidomastoid muscle; Trapezius; neck pain musculoskeletal
MeSH Terms: conditions — Neck Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled trial. Total 60 patients will be recruited, 30 in each group that includes 6 patients as a dropout in both groups. There will be one interventional group and one control group. Treatment will be allocated using a random number sheet generated by SPSS software version 23. Participants are assigned to one of two groups in parallel for the duration of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes assessor involved in the clinical trial will be prevented from having knowledge of the interventions assigned to individual participants. Participants will also be masked as both treatments are almost similar.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Intervention) (Experimental): To start Progressive Muscle Relaxation Technique with deep breathing, individuals will be trained to sit in a comfortable position with or without eyes opening. It will involve relaxing neck muscles through a two-step process. First, participants will be commanded to tense the particular SCM and upper trapezius muscle by active contraction along with deep breathing (deeply and slowly inhaling through the nose). Then, they will be commanded to squeeze the muscles as hard as they can, holding for 5-10 seconds, after that employees will be asked to relax the muscle for 10-15 seconds while relaxing the muscle employees will be asked to exhale slowly through the mouth (5 repetitions for each side). Intervention will be given for 30 minutes for 6 days a week for 2 weeks.
  Interventions: Other: Progressive Muscle Relaxation Technique
- Group B (Control) (Active Comparator): Muscle Energy Technique with deep breathing
  * Trapezius Muscle: The therapist will position the patient supine, supporting the back of the patient's head with one hand and placing the other on the clavicle. The head will be bent forward, rotated, and bent toward the same side to test for flexibility, and then brought midway between the initial and fully rotated positions. The patient will breathe in, hold their breath, and perform isometric (20% of max force) while the therapist provides resistance for 6-7 seconds, followed by a stretch during exhalation, to be repeated 3-4 times.
  * Sternocleidomastoid Muscle: The patient will be supine with a cushion under the shoulder, tilting the head slightly back. The therapist will place one hand on the mastoid and the other on the sternum. The patient will rotate the head to the opposite side, lift it while holding breath while the therapist provides resistance for 6-7 second
  Interventions: Other: Muscle Energy Technique

INTERVENTIONS:
Other: Progressive Muscle Relaxation Technique — Progressive Muscle Relaxation (PMR) is a relaxation technique that involves systematically tensing and then relaxing different muscle groups in the body to reduce physical tension and stress. Developed by Edmund Jacobson in the 1930s, PMR aims to promote deep relaxation by increasing awareness of muscle tension and learning to release it. The technique is typically performed in a quiet environment, starting from the feet and progressing upward or vice versa. It is commonly used for stress management, pain relief, anxiety reduction, and improving overall well-being.
  Arms: Group A (Intervention)
Other: Muscle Energy Technique — Muscle Energy Technique (MET) is a manual therapy approach that uses the patient's voluntary muscle contractions against a controlled resistance provided by the therapist to improve musculoskeletal function. It is commonly used to lengthen shortened muscles, improve joint mobility, and reduce pain. MET works by engaging the target muscles in an isometric or isotonic contraction, followed by a relaxation phase, allowing for a greater stretch or repositioning of the joint. It is frequently used in physiotherapy for conditions such as muscle tightness, joint restrictions, and postural imbalances.
  Arms: Group B (Control)

SUMMARY:
The objective of this randomized controlled trial is to assess the potential effectiveness of Progressive muscle relaxation technique (PMRT) vs Muscle energy technique (MET) as an intervention for releasing trigger points in SCM and upper trapezius in prolonged computer users. The study will be conducted in a workplace setting, where desk-type computer users are expected to regularly engage in their professional activities for ≥ 6 hours throughout the day, intermittently. This study will be conducted at the Outpatient Physiotherapy department of Sindh Institute of Physical Medicine and Rehabilitation, Karachi among 60 patients with nonspecific chronic neck pain on the basis of non-probability purposive sample technique. After taking informed consent, all participants will be randomly allocated into two groups through a investigator (blinded) the same investigator will be screening the individuals, doing baseline assessment, and post treatment assessment while another investigator will be providing intervention. Group 1 will receive Progressive muscle relaxation technique while Group 2 will receive Muscle Energy Technique on sternocleidomastoid and upper trapezius bilaterally. Patients will also be blinded. A total of 12 sessions will be provided. Outcomes will be assessed at baseline and post treatment after 2 weeks intervention.

ELIGIBILITY:
Inclusion Criteria:

* Persons using computer more than 6 hours throughout the day, intermittently both genders.
* Age between 20-45.
* Hypertonicity of trapezius muscle and SCM muscle. Specifically, those workers have neck pain and stiffness (including trouble tilting or turning head). Patients who reported small tightening and spasm at the posterior aspect of their neck are included, also associated with more diffuse neck pain patterns that included the following: headache, (upper back, neck and shoulder pain) numbness/ tingling in the hand/arm.
* Pain intensity of 2 on the NRS and presence of at least one latent trigger point in a taut band in the neck region.

Exclusion Criteria:

* Recent trauma to the cervical region
* Exclusion criteria based on with any serious pathology such as specific neck pain due to disc prolapsed, tumor of cervical spine, whiplash injury, cervical fractures, Cervicogenic headache, and any neurological signs consistent with nerve root compression

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain on Numeric Rating Scale | Baseline and week 2
  On a scale of 0 to 10, with 0 being no pain and 10 being the worst pain imaginable. Individuals will be asked to rate the pain. Increase in number suggests increase in pain and decrease in number suggests decrease in pain.
Change in disability on the Neck Pain Disability Index Scale | Baseline and week 2
  The questionnaire, consists of 10 sections with scores ranging from 0 to 5, has demonstrated validity and reliability. The percentage of disability score will be calculated, where item scores range from 0 (no limitation) to 5 (major activity limitation), and the total score is a sum of the item scores (possible range 0 (no pain) - 50 (maximal pain)). A score of less than 4 indicates no disability; 5-14 mild disability, 15-24 moderate disability and 25-34 severe disability. A score of above 35 indicate complete perceived disability. The patient will rate each section based on their level of difficulty due to neck pain. Increase in score suggests increase in disability and decrease in score suggests decrease in disability.

SECONDARY OUTCOMES:
Change in Range of Motion on the Goniometer | Baseline and week 2
  A goniometer, a tool used to measure joint angles, is used to assess range of motion, which is the degree of movement a joint can achieve. Goniometry, the measurement of joint angles. Increase in scores suggests increase in range of motion.
Change from baseline in head posture on plumb line | Baseline and week 2
  A plumb line is a simple tool to check posture by comparing head and shoulder alignment. Landmarks: Mastoid process & auditory meatus (ear canal). Any forward head posture is noted if the tragus (ear) moves ahead of the plumb line. Measured in inches while standing or sitting. Increase in inches suggests increase and decrease suggests decrease in forward head posture.

CONTACTS AND LOCATIONS:
Overall Officials: Syeda Waniya Riaz, PhD (scholar), MSAPT, DPT, Principal Investigator — IQRA University
Locations (1):
- Sindh Institute of Physical Medicine and Rehabilitation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
The investigators will publish the results in academic journals. The study data will be shared through multiple channels. We aim to make our findings accessible to researchers and potential collaborators with an interest in physical medicine, rehabilitation, and chronic neck pain.

REFERENCES:
- [Background] Ramasamy S, Panneerselvam S, Govindharaj P, Kumar A, Nayak R. Progressive muscle relaxation technique on anxiety and depression among persons affected by leprosy. J Exerc Rehabil. 2018 Jun 30;14(3):375-381. doi: 10.12965/jer.1836158.079. eCollection 2018 Jun. PMID 30018921
- [Background] Batool A, Soomro RR, Baig AAM. Comparing the effects of neck stabilization exercises versus dynamic exercises among patients having nonspecific neck pain with forward head posture: a randomized clinical trial. BMC Musculoskelet Disord. 2024 Sep 4;25(1):707. doi: 10.1186/s12891-024-07749-8. PMID 39232708
- [Background] Sukari AAA, Singh S, Bohari MH, Idris Z, Ghani ARI, Abdullah JM. Examining the Range of Motion of the Cervical Spine: Utilising Different Bedside Instruments. Malays J Med Sci. 2021 Apr;28(2):100-105. doi: 10.21315/mjms2021.28.2.9. Epub 2021 Apr 21. PMID 33958964
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Bielewicz J, Daniluk B, Kamieniak P. VAS and NRS, Same or Different? Are Visual Analog Scale Values and Numerical Rating Scale Equally Viable Tools for Assessing Patients after Microdiscectomy? Pain Res Manag. 2022 Mar 29;2022:5337483. doi: 10.1155/2022/5337483. eCollection 2022. PMID 35391853
- [Background] Rezaeian T, Mosallanezhad Z, Nourbakhsh MR, Noroozi M, Sajedi F. Effects of Dry Needling Technique Into Trigger Points of the Sternocleidomastoid Muscle in Migraine Headache: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2020 Dec;99(12):1129-1137. doi: 10.1097/PHM.0000000000001504. PMID 32544109
- [Background] Pathan NM, Thakur S, Kadam K, Lohade S, Chandak N. Immediate effects of positional release therapy and manual trigger point release on neck pain and range of motion in computer users with upper trapezitis. J Family Med Prim Care. 2021 Aug;10(8):2839-2844. doi: 10.4103/jfmpc.jfmpc_1608_20. Epub 2021 Aug 27. PMID 34660415
- [Background] Khan ZK, Ahmed SI, Baig AAM, Farooqui WA. Effect of post-isometric relaxation versus myofascial release therapy on pain, functional disability, rom and qol in the management of non-specific neck pain: a randomized controlled trial. BMC Musculoskelet Disord. 2022 Jun 13;23(1):567. doi: 10.1186/s12891-022-05516-1. PMID 35698187
- [Background] Lauche R, Materdey S, Cramer H, Haller H, Stange R, Dobos G, Rampp T. Effectiveness of home-based cupping massage compared to progressive muscle relaxation in patients with chronic neck pain--a randomized controlled trial. PLoS One. 2013 Jun 7;8(6):e65378. doi: 10.1371/journal.pone.0065378. Print 2013. PMID 23762355
- [Background] Sbardella S, La Russa C, Bernetti A, Mangone M, Guarnera A, Pezzi L, Paoloni M, Agostini F, Santilli V, Saggini R, Paolucci T. Muscle Energy Technique in the Rehabilitative Treatment for Acute and Chronic Non-Specific Neck Pain: A Systematic Review. Healthcare (Basel). 2021 Jun 17;9(6):746. doi: 10.3390/healthcare9060746. PMID 34204590
- [Background] Loh EW, Shih HF, Lin CK, Huang TW. Effect of progressive muscle relaxation on postoperative pain, fatigue, and vital signs in patients with head and neck cancers: A randomized controlled trial. Patient Educ Couns. 2022 Jul;105(7):2151-2157. doi: 10.1016/j.pec.2021.10.034. Epub 2021 Nov 3. PMID 34785078
- [Background] Liu K, Chen Y, Wu D, Lin R, Wang Z, Pan L. Effects of progressive muscle relaxation on anxiety and sleep quality in patients with COVID-19. Complement Ther Clin Pract. 2020 May;39:101132. doi: 10.1016/j.ctcp.2020.101132. Epub 2020 Mar 6. PMID 32379667
- [Background] Vambheim SM, Kyllo TM, Hegland S, Bystad M. Relaxation techniques as an intervention for chronic pain: A systematic review of randomized controlled trials. Heliyon. 2021 Aug 20;7(8):e07837. doi: 10.1016/j.heliyon.2021.e07837. eCollection 2021 Aug. PMID 34485731
- [Background] Toussaint L, Nguyen QA, Roettger C, Dixon K, Offenbacher M, Kohls N, Hirsch J, Sirois F. Effectiveness of Progressive Muscle Relaxation, Deep Breathing, and Guided Imagery in Promoting Psychological and Physiological States of Relaxation. Evid Based Complement Alternat Med. 2021 Jul 2;2021:5924040. doi: 10.1155/2021/5924040. eCollection 2021. PMID 34306146
- [Background] Jun D, Johnston V, McPhail SM, O'Leary S. A Longitudinal Evaluation of Risk Factors and Interactions for the Development of Nonspecific Neck Pain in Office Workers in Two Cultures. Hum Factors. 2021 Jun;63(4):663-683. doi: 10.1177/0018720820904231. Epub 2020 Mar 2. PMID 32119582
- [Background] Kashyap R, Iqbal A, Alghadir AH. Controlled intervention to compare the efficacies of manual pressure release and the muscle energy technique for treating mechanical neck pain due to upper trapezius trigger points. J Pain Res. 2018 Dec 12;11:3151-3160. doi: 10.2147/JPR.S172711. eCollection 2018. PMID 30588067
- [Background] Shah JP, Thaker N, Heimur J, Aredo JV, Sikdar S, Gerber L. Myofascial Trigger Points Then and Now: A Historical and Scientific Perspective. PM R. 2015 Jul;7(7):746-761. doi: 10.1016/j.pmrj.2015.01.024. Epub 2015 Feb 24. PMID 25724849
- [Background] Sabeen F, Bashir MS, Hussain SI, Ehsan S. Prevalance of neck pain in computer users. Ann King Edw Med Univ. 2013;19(2):137-43.
- [Background] Chakraborty S, Chatterjee DSS, Basu M, et al. A Study on Work Related Neck Pain among Bank Employees in Kolkata, India. Int J Contemp Med Res. 2020;7(6):F1-8.
- [Background] Park J, Kim H, Kim KW, Cho JH, Chung WS, Song MY. Bibliometric Analysis of Research Trends on Acupuncture for Neck Pain Treatment Over the Past 20 Years. J Pain Res. 2021 Oct 12;14:3207-3221. doi: 10.2147/JPR.S331514. eCollection 2021. PMID 34675647
- [Background] Bodin T, Berglund K, Forsman M. Activity in neck-shoulder and lower arm muscles during computer and smartphone work. Int J Ind Ergon. 2019;74:102870.
- [Background] Oha K, Animagi L, Paasuke M, Coggon D, Merisalu E. Individual and work-related risk factors for musculoskeletal pain: a cross-sectional study among Estonian computer users. BMC Musculoskelet Disord. 2014 May 28;15:181. doi: 10.1186/1471-2474-15-181. PMID 24884911
- [Background] Marker RJ, Balter JE, Nofsinger ML, Anton D, Fethke NB, Maluf KS. Upper trapezius muscle activity in healthy office workers: reliability and sensitivity of occupational exposure measures to differences in sex and hand dominance. Ergonomics. 2016 Sep;59(9):1205-14. doi: 10.1080/00140139.2015.1130860. Epub 2016 Feb 28. PMID 26924036
- See also: Related Info — https://www.researchgate.net/publication/284168992_Prevalance_of_Neck_Pain_in_Computer_Users
- See also: Stress effects on the body [Internet]. American Psychological Association — https://www.apa.org/topics/stress/body
- See also: Jacobson, E. Progressive relaxation. Chicago: University of Chicago Press. 1929. — https://www.scirp.org/reference/referencespapers?referenceid=1146522
- See also: Progressive muscle relaxation: Benefits, techniques, and more [Internet]. MediLexicon International. — https://www.medicalnewstoday.com/articles/progressive-muscle-relaxation-pmr
- See also: Norelli SK, Long A, Krepps JM. Relaxation Techniques. StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing. 2021. — https://www.ncbi.nlm.nih.gov/books/NBK513238/